CLINICAL TRIAL: NCT03754140
Title: Intralesional Sclerosant for in Transit and Cutaneous Melanoma Metastases
Acronym: INTRANS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to identify eligible patients within planned timeframe
Sponsor: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/18/RPAH 621
Record Dates: First submitted 2018-10-31; First posted 2018-11-27 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Melanoma; In-Transit Metastasis of Cutaneous Melanoma
Keywords: Sclerosant; Polidocanol
MeSH Terms: conditions — Melanoma | interventions — Polidocanol

STUDY DESIGN:
Intervention Model Description: Open label, single arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polidocanol Injection (Experimental): Polidocanol (3%) 0.1ml intralesional injection per 10mm diameter lesion
  Interventions: Drug: Polidocanol Injection

INTERVENTIONS:
Drug: Polidocanol Injection — Sclerotic agent
  Other Names: Aethoxysklerol

SUMMARY:
There is currently an urgent need for low cost and well tolerated intralesional agents for the management of in transit and cutaneous melanoma metastases that are unsuitable for, or resistant to, other therapies. This pilot study will determine whether intralesional injections of the sclerosant polidocanol into intransit and cutaneous melanoma lesions shows promise for efficacy, safety and ease of use that will enable this inexpensive and widely available agent to undergo further evaluation.

DETAILED DESCRIPTION:
Many patients with metastatic melanoma have in transit and other cutaneous metastases. Untreated, these lesions become eroded, haemorrhagic and symptomatic. When systemic therapy is not warranted, has failed or is not tolerated for in transit disease, and when surgery is not feasible or appropriate, other local treatments are needed. Current options include isolated limb infusion for bulky limb disease, topical immunotherapy with contact sensitisers and imiqiuimod for superficial, nonbulky disease or radiation therapy. Intralesional (IL) agents such as Rose Bengal (PV-10, Provectus) and Talimogene laherparepvec (T-Vec, Amgen) have been used for patients with limited numbers of cutaneous metastases with reported overall response rates of 51% and 26% respectively. It is thought that these IL agents can incite regional or even systemic anti-tumour immune responses, thus providing benefit beyond the individual injected lesions. Use of PV-10, which is not an intrinsic immune modulator, was associated with regression of untreated bystander lesions in 27% of patients.

T-Vec is not currently available as a subsidised product in Australia and PV-10 is not currently accessible outside of dual-agent systemic/IL clinical trials. Intralesional injection of the antimetabolites 5-fluorouracil and methotrexate has been used successfully for the treatment of cutaneous squamous cell carcinoma, but the efficacy of these agents in melanoma is unknown. Importantly, the investigator's in transit melanoma patients usually have multiple, often very numerous lesions, making IL injection with adequate volumes of antimetabolites difficult without significant risk of systemic haematologic, hepatic and renal side effects.

Hence there is currently an urgent need for tolerable, low cost and accessible intralesional therapies for in transit and cutaneous melanoma metastases.

This study aims to evaluate the efficacy and tolerability of intralesional therapy with the sclerosant polidocanol for treatment of in transit and cutaneously metastatic melanoma unsuitable for other therapies.

Intravascularly injected sclerosants have a long history of safe and effective use in the treatment of varicose veins. Sclerosants have also been used intralesionally for the treatment of cutaneous lesions such as squamous cell carcinoma, pyogenic granulomas, Kaposi sarcoma and angiomas. They are inexpensive, readily accessible and can be easily administered in the clinic to multiple metastases. By inciting cell death within melanoma metastases in the skin, they may also incite anti-tumour immune responses in untreated bystander lesions, as is observed with IL PV-10 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed in transit and/or cutaneous melanoma metastases unsuitable for, or with progressive disease despite systemic, surgical, intra-arterial, topical or radiation therapies
* A minimum of 2 accessible lesions

Exclusion Criteria:

* Periocular lesions
* Severe renal impairment defined as an estimated glomerular filtration rate <20ml/min/1.73sqm
* Sever liver function abnormality defined as aspartate aminotransferase and / or alanine aminotransferase > 3 x upper limit of normal and / or bilirubin > 1.5 x upper limit of normal
* known hypersensitivity to polidocanol or its exipients
* Patients unavailble for the full study duration (of a 4 week screening period and 8 week treatment period) because of general frailty, geographical or social reasons
* Pregnant or breast feeding female patients
* Patients receiving topical or radiation therapy to the in transit and / or cutaneous lesions within 4 weeks of planned start of study treatment (patients receiving current systemic immunotherapy which is deemed appropriate to continue, despite progression of disease in the skin, in order to reduce the likelihood of visceral metastases are eligible)
* Patients receiving sclerosants for other indications within 4 weeks of planned start of study treatment or during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of interlesional polidocanol injection assessed by the size of in transit melanoma metastases after treatment | 8 weeks
  Proportion of patients with a complete response (complete disappearance of treated lesions), partial response (a 25% or more reduction in size of treated lesions), stable disease (a 0 to 24% reduction in size of treated lesions) or disease progression (any increase in size of treated lesions)

SECONDARY OUTCOMES:
Incidence of treatment related adverse events | 8 weeks
  Treatment related adverse events using the CTCAE version 4 terms and grading.
Bystander treatment effect on untreated intransit melanoma metastases | 8 weeks
  Proportion of patients with a complete response (complete disappearance of untreated lesions), partial response (a 25% or more reduction in size of untreated lesions), stable disease (a 0 to 24% reduction in size of untreated lesions) or disease progression (any increase in size of untreated lesions)
Bystander treatment effect on the proportion of tumour infiltrating immune markers in treated and untreated melanoma lesions | 8 weeks
  The proportion (%) of tumour-infiltrating immune markers: CD4, CD8 and FoxP3 T cell markers, CD20 (B cell), CD16 and CD56 Natural Killer (NK) cell markers, Ki67 marker of proliferation, CD31 (endothelial cells) and CD68 and CD163 (macrophages) detected at baseline and 1 week after intralesional injection by immunohistochemistry. The same analysis will be undertaken in a minimuim of one untreated lesion detected at baseline and at anytime between 1 and 8 weeks. Change in the proportion (%) of immune markers will be ,made within each lesion and between each lesion.
Bystander treatment effect on tumour viabilty in treated and untreated melanoma lesions | 8 weeks
  The proportion of residual non-necrotic melanoma cells detected histolologcally in treated and untreated lesions one week after intralesional injection.

CONTACTS AND LOCATIONS:
Overall Officials: Diona Damian, Study Director — Royal Prince Alfred Hospital, Sydney, Australia
Locations (1):
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No